CLINICAL TRIAL: NCT05279339
Title: The Relationship Between Subjective and Objective Changes in Muscle-stiffness
Brief Title: Subjective and Objective Changes in Muscle-stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Steffan Wittrup Christensen, Associate Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AAU031-1004903
Record Dates: First submitted 2022-02-16; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Healthy; Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will not perform any exercise
- Exercise (Experimental): Participants will perform an exercise recommended for preventing neck and shoulder pain
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Upper limb exercises using an elastic band.
  Arms: Exercise

SUMMARY:
The purpose of this study is to investigate muscle stiffness in relation to delayed on-set muscle soreness following exercise and to investigate how well the change in muscle stiffness correlates with the subjective experienced degree of stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 18-80
* Able to speak, read and understand Danish and/or English

Exclusion Criteria:

* Have performed resistance training on a regular basis during the past month
* Experience of delayed onset muscle soreness (DOMS) during the last two weeks leading up to the first test session
* Current use of analgesics
* Any current neurological, musculoskeletal or mental illnesses that could interfere with the results.
* Pregnancy
* Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscle stiffness (change) - Shear wave | Day1,Day 2 and Day7
  Muscle stiffness measured by ultrasound using shear wave elastography

SECONDARY OUTCOMES:
Muscle stiffness (change) - Self-reported | Day1,Day 2 and Day7
  Self-reported muscle stiffness: Measured on a NRS scale (0-10), where 0 = not stiff at all, 10 is maximal stiffness
Muscle stiffness (change) - Myotonometry | Day1,Day 2 and Day7
  Muscle stiffness measured by Myotonometry
Muscle stiffness (change)- Palpation | Day1,Day 2 and Day7
  Muscle palpation: Reported using a 5-point Likert: 1 = very low muscle stiffness and 5 = very high muscle stiffness

OTHER OUTCOMES:
Muscle thickness | Day1,Day 2 and Day7
  Muscle thickness measured by ultrasound
Muscle soreness | Day1,Day 2 and Day7
  Self-reported muscle soreness: Measured on a NRS scale (0-10), where 0 = not sore at all, 10 is maximal soreness
Neck disability | Day1,Day 2 and Day7
  The NDI is questionnaire investigating neck pain and disability: Scores range from 0 to 50. Higher score represent worse disability
Shoulder disability | Day1,Day 2 and Day7
  SPADI is a 13-item questionnaire investigating shoulder pain and disability: Scores range from 0 to 130. Higher score represent worse disability

CONTACTS AND LOCATIONS:
Overall Officials: Steffan WM Christensen, PhD, Principal Investigator — Aalborg University
Locations (1):
- Dept. Of Health Science and Technology, Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No